CLINICAL TRIAL: NCT04494633
Title: Summative Assessment of the BurntOut 3D Simulation With Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Tools, Inc. (Industry)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 271330; R44AA026474 (NIH)
Record Dates: First submitted 2020-07-10; First posted 2020-07-31 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Burnout, Student; Alcohol; Harmful Use; Quality of Life; Depression; Resilience; Drug Use; Burnout, Professional
MeSH Terms: conditions — Burnout, Psychological; Depression; Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants completed the pre-assessments, used the intervention, waited 2-4 weeks, and then completed the assessments again.
  Interventions: Other: Clinical Encounters Medical School 3D Simulation
- Wait Group (No Intervention): Participants completed the pre-assessments, waited 2-4 weeks, and completed the assessments again.

INTERVENTIONS:
Other: Clinical Encounters Medical School 3D Simulation — A 3D simulation related to coping with the stresses of medical school and burnout.
  Arms: Intervention

SUMMARY:
Burnout is a common problem for medical students and is associated with stress-related health problems and also potentially affects the quality of care delivered to their patients. Among the health problems commonly associated with burnout are substance use problems, and alcohol is the substance most often misused. The purpose of the evaluation is to document whether an educational intervention incorporating aspects of virtual reality (VR) via a 3D online simulation experience prevents or improves the primary endpoint of burnout and the secondary endpoints of burnout-related factors in medical students. The investigators will also will evaluate student satisfaction with the intervention to determine if it meets our standard of success. The hypothesis is that the intervention will improve the primary clinical endpoint of burnout from pre-intervention to post-intervention as measured by the Maslach Burnout Inventory, a validated inventory that is widely used to measure burnout. The related factors that will be measured as secondary clinical endpoints include quality of life, substance use (alcohol and drugs), depression, and resilience. Due to evidence that these endpoints are linked to burnout, the investigators also hypothesize that the measures will improve pre- to post-intervention. Satisfaction of the target audience after completing the simulation intervention will also be evaluated. The evaluation will be prior to and after use of the simulation by medical student participants, using a pre-/post intervention, wait-list control, parallel design.

DETAILED DESCRIPTION:
The investigators used a pre-/post-intervention design with wait-list controls who were able to use the intervention after the study, if they chose. The investigators recruited and enrolled 73 medical students. The number of participants selected is based on a power analysis of the design and experience of low dropout rate with this target audience; to reach a medium effect size the investigators plan for a final sample size of 68 medical students and 63 actually completed the study. During the intervention phase of the study, intervention group students 1) Completed the simulation experience: an interactive online simulation, interactive online case stories, and resilience-building activities (taking around 2 hours over a period of less than 2 weeks); and 2) Completed pre- assessments and 2-4 week post-assessments (each taking <1 hour). Controls completing pre-assessments and repeated the pre assessments after a 2 to 4 week wait period. The investigators screened for and excluded students with severe depression and suicidality but none needed to be excluded for this reason. The primary clinical endpoint was burnout as measured by the Maslach Burnout Inventory. Secondary endpoints were measured via adaptations of the following assessments: Alcohol Use Disorders Identification Test (AUDIT-C/AUDIT) for alcohol use disorder, Patient Health Questionaire (PHQ2/PHQ9) to screen for depression, Connor-Davidson Resilience Scale © (CD-RISC 2) for resiliency, two drug question screening for drug use, and Medical Student Quality of Life (MSQoL9). Control participants were invited to engage in the intervention after completing the study, that is, after completing their 2nd set of assessments. There were no adverse events.

ELIGIBILITY:
Inclusion Criteria:

* US Medical students in years 2-4
* Has access to a computer with Internet access

Exclusion Criteria:

--Self report of active symptoms of major depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary P Metcalf, PhD, Principal Investigator — Clinical Tools, Inc.
Locations (1):
- Clinical Tools, Inc., Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from lists of medical student emails at multiple US medical schools. Recruitment and the study started on the same date and continued until sufficient students had started plus allowance for expected dropout rate.
Groups:
- Wait Group: Participants will complete the pre-assessments, wait 2-4 weeks, and complete the assessments again. They were then given the option to use the intervention.
- Intervention: Participants will complete the pre-assessments, use the intervention, wait 2-4 weeks, and complete the assessment a 2nd time.
Period: Overall Study
Arm/Group | Wait Group | Intervention
Started | 35 | 38
Completed | 29 | 34
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 5 | 3
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Wait Group: Participants will complete the pre-assessments, wait 2-4 weeks, complete the assessments, use the intervention, complete the assessment a 3/final time.
  Clinical Encounters Medical School VR Simulation: A VR simulation related to coping with the stresses of medical school and burnout.
- Intervention: Participants will complete the pre-assessments, use the intervention, complete the assessments, wait 2-4 weeks, and complete the assessment a 3/final time.
  Clinical Encounters Medical School VR Simulation: A VR simulation related to coping with the stresses of medical school and burnout.
- Total: Total of all reporting groups
Arm/Group | Wait Group | Intervention | Total
Number analyzed (Participants) | 29 | 34 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 34 | 63
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 26 | 37
  Male | 18 | 8 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian | 0 | 0 | 0
  Asian/PI | 12 | 9 | 21
  Black or African American | 1 | 3 | 4
  More than One Race | 4 | 3 | 7
  Other | 1 | 2 | 3
  Prefer Not To Answer | 1 | 0 | 1
  Caucasian/White | 10 | 17 | 27
Region of Enrollment [Number; unit: participants]
  United States | 29 | 34 | 63
Maslach Burnout Inventory (MBI) (modified) [Mean (Standard Deviation); unit: units on a scale] — Measure of burnout. Measure modified to eliminate questions that are not relevant for medical student burnout.
  Value reported is mean total score. 16 questions. Range for total score: 0 to 96. Higher score means worse outcome, greater burnout. Results modified in the analysis so that a higher score for all questions means more burnout.
  7 point Likert scale: Never=0; A few times a year or less=1; Once a month or less=2; A few times a month=3; Once a week=4; A few times a week=5; Every day=6
  units on a scale | 41.34 (16.09) | 41.44 (15.22) | 41.40 (15.5)
Alcohol Use Disorders Identification Test - Concise (AUDIT-C) [Mean (Standard Deviation); unit: units on a scale] — Value reported is mean total score. 3 questions Range for total Score: 0-12. Higher score means worse outcome, greater use of alcohol.
  5 point Likert scale: Question 1. 0=Never; 1=Monthly or Less; 2=2-4 times a month; 3=2-3 times a week; 4=4 or more times a week Question 2. 0=N/A; 0=1 or 2; 1=3 to 4; 2=5 to 6; 3=7 to 9; 4=10 or more Question 3. 0=Never; 1=Less than monthly; 2=Monthly; 3=Weekly; 4=Daily or almost daily
  units on a scale | 3.07 (1.79) | 2.71 (1.49) | 2.87 (1.63)
Patient Health Questionnaire (PHQ) - modified [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire-9 screen for depression, selected questions used. Value reported is mean total score. 6 questions Range per total score 0-24. Higher values mean more severe depression. Likert scale 1st 5 questions: Not at all (0 days)=0; Several days (1-6 days)=1; More than half the days (7+ days)=2; Nearly every day (~14 days)=3; 6th question scale: Not at all difficult=0; Not very difficult=1; Difficult=2; Very difficult=3
  units on a scale | 4.55 (3.86) | 3.85 (3.43) | 4.17 (3.62)
Connor-Davidson Resilience Scale (CD-RISC) [Mean (Standard Deviation); unit: units on a scale] — Selected questions from the Connor Davidson-Resilience scale. Value entered is mean total score. 2 questions evaluation of resiliency, Range per total survey score 0-8. Higher scores mean better outcome, greater resilience. Likert scale: Not true at all=0; Rarely true=1; Sometimes true=2; Often true=3; True nearly all the time=4.
  units on a scale | 5.83 (1.47) | 6.27 (1.56) | 6.06 (1.52)
National Institute on Drug Abuse (NIDA) Quick Screen [Mean (Standard Deviation); unit: units on a scale] — Screen for use of drugs. (Modified to add "Other than cannabis to 2nd question on illegal drugs)" Value reported is mean total score. 2 questions Higher value means worse outcome, greater drug use. Range per question (1-5), per total score (1-15): Scale: Never=1; Monthly or less=2; 2-4 times a month=3; 2-3 times a week=4; 4 or more times a week=5
  units on a scale | 2.28 (0.88) | 2.12 (0.73) | 2.19 (0.80)
Medical Student Quality of Life [Mean (Standard Deviation); unit: units on a scale] — Measures exhaustion and happiness. Value reported is mean total score (SD). 5 questions (Range per total score 1-25) Modified so that higher scores mean better outcomes, for all questions, ie, more energy and happiness and less exhaustion. Scale per question: Never=1, A little of the time=2, A good bit of the time=3, Most of the time=4, All of the time=5
  units on a scale | 15.07 (3.29) | 15.32 (2.68) | 15.21 (2.96)

OUTCOME MEASURES:

1. Primary Outcome: Burnout Change
Description: Burnout was measured using the Maslach Burnout Inventory (modified). This scale uses items to assess emotional exhaustion, and depersonalization, and measure the sense of personal accomplishment. Selected items were used to make it relevant to medical students experience. It was modified so that for all questions, higher scores indicate higher, and thus more problematic, levels of burnout.
  A decrease means an improvement; lower values mean more improvement. A positive change means worsening; higher values mean more worsening.
  Range: Minimum total value 0, Maximum total value 96.
  The Outcome Measure is the amount of Burnout Change from baseline (evaluation point #1) to evaluation point #2. Burnout Change is calculated for the intervention group pre intervention and 2 weeks post intervention (case) and pre intervention and after a 2 week waiting period for the Wait Group (Control) .
  See Baseline for more details.
Time Frame: 1 months
Population: Medical students in the US
Measure: Mean (Standard Deviation); unit: change in score on a scale
Groups:
- Intervention: Participants will complete the pre-assessments, use the intervention, wait 2-4 weeks, and complete the assessment again.
  Clinical Encounters Medical School VR Simulation: A VR simulation related to coping with the stresses of medical school and burnout.
Arm/Group | Wait Group | Intervention
Number analyzed (Participants) | 29 | 34
change in score on a scale | 0.06 (0.24) | 0.05 (0.51)
Statistical Analysis 1: Comparison: Wait Group vs Intervention; Test type: Superiority; p = 0.482314, t-test, 2 sided; The change for each group was analyzed using a 2-tailed, unpaired, independent means, t-test with 61 degrees of freedom

2. Secondary Outcome: Alcohol Use Change
Description: Alcohol use was measured using the Alcohol Use Disorders Identification Test - Concise, (AUDIT-C). This instrument is a screening tool to identify users who are hazardous drinkers or who have active alcohol use disorder.
  Higher scores= greater frequency or amount of alcohol use or misuse
  Range: Minimum value: 0, Maximum value 12. High scores indicate worse outcomes. A score of over 4 for men, and over 3 for women is considered a positive screen for alcohol misuse. Higher scores suggest a higher likelihood that alcohol use is negatively impacting the person's health and safety.
  The Outcome Measure is the amount of Alcohol Use Change from baseline (evaluation point #1) to evaluation point #2. Alcohol Use Change was calculated for the intervention group pre intervention and 2 weeks post intervention (case) and pre intervention and after a 2 week waiting period for the Wait Group (Control) .
Time Frame: 1 months
Population: Medical student participants
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Wait Group | Intervention
Number analyzed (Participants) | 29 | 34
change in score on a scale | -0.03 (0.78) | 0 (.95)
Statistical Analysis 1: Comparison: Wait Group vs Intervention; Test type: Superiority; p = .876964, t-test, 2 sided; The change for each group was analyzed using a 2-tailed, unpaired, independent means, t test with 61 degrees of freedom

3. Secondary Outcome: Depression Change
Description: Depression was measured using the Patient Health Questionaire, PHQ-9 (modified to 6 questions). The PHQ is a screen where respondents indicate how often the respondent has experienced depressed mood and anhedonia over the prior two weeks. Selected questions (6) were used.
  Range: Minimum score: 0, Maximum score18. High scores indicate worse outcomes.
  The Outcome Measure is the amount of Depression Change from baseline (evaluation point #1) to evaluation point #2. Depression Change is calculated for the intervention group pre intervention and 2 weeks post intervention (case) and pre intervention and after a 2 week waiting period for the Wait Group (Control).
  See Baseline for more details
Time Frame: 1 months
Population: Medical student participants
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Wait Group | Intervention
Number analyzed (Participants) | 29 | 34
change in score on a scale | -0.28 (1.96) | -0.53 (2.57)
Statistical Analysis 1: Comparison: Wait Group vs Intervention; Test type: Superiority; p = .66602, t-test, 2 sided; The change for each group was analyzed using a 2-tailed, unpaired, independent means, with 61 degrees of freedom

4. Secondary Outcome: Resilience Change
Description: Resilience was measured via the Connor-Davidson Resilience Scale - modified to use 2 questions from the scale.
  Range: Minimum score: 0, Maximum score: 8.
  An increase means an improvement and higher scores mean better outcomes. A decrease means worsening; and lower values mean worse outcomes.
  The Outcome Measure is the amount of Resilience Change from baseline (evaluation point #1) to evaluation point #2. Resilience Change was calculated for the intervention group pre intervention and 2 weeks post intervention (case) and pre intervention and after a 2 week waiting period for the Wait Group (Control).
  See Baseline for more details.
Time Frame: 1 months
Population: Medical student participants
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | Wait Group | Intervention
Number analyzed (Participants) | 29 | 34
Change in score on a scale | 0.1 (1.21) | 6.26 (1.38)
Statistical Analysis 1: Comparison: Wait Group vs Intervention; Test type: Superiority; p = .726421, t-test, 2 sided; Two-tailed unpaired t test comparing change for control (Pre to 2 weeks later) to case (Pre- to 2 weeks post) with 61 degrees of freedom

5. Secondary Outcome: Drug Use Change
Description: Drug use in the recent past was measured via the National Institute for Drug Abuse-Modified Alcohol, Smoking and Substance Involvement Screening Test (modified to use 2 questions from this scale).
  Range: Minimum 0, Maximum score 10.
  High scores indicate more drug use and an increase means worse outcomes. Low scores mean less drug use and a decrease means better outcomes.
  The Outcome Measure is the amount of Drug Use Change from baseline (evaluation point #1) to evaluation point #2. Drug Use Change is calculated for the intervention group pre intervention and 2 weeks post intervention (case) and pre intervention and after a 2 week waiting period for the Wait Group (Control).
  See Baseline for more details.
Time Frame: 1 months
Population: Medical students
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Wait Group | Intervention
Number analyzed (Participants) | 29 | 34
change in score on a scale | -0.07 (0.88) | -.09 (0.38)
Statistical Analysis 1: Comparison: Wait Group vs Intervention; Test type: Superiority; p = 0.908468, t-test, 2 sided; The statistical test used was a 2 tailed, unpaired t test with 61 degrees of freedom

6. Secondary Outcome: Happiness and Exhaustion (Quality of Life)
Description: Happiness and Exhaustion (Quality of Life) were measured using the Medical Student Quality of Life Questionnaire with Nine Items (MSQoL9). The MSQoL is a linear self-assessment analog scale. It was modified to use only 5 of the questions from the scale that are on the domains of exhaustion and general happiness.
  Range for total score on the 5 questions: 1-25
  Greater increase in scores means improvement; High scores indicate better outcomes. The analysis was modified so that high scores indicate a better quality of life for all questions.
  The Outcome Measure is the amount of Happiness and Exhaustion (Quality of Life) Change from baseline (evaluation point #1) to evaluation point #2. Happiness and Exhaustion (Quality of Life) Change was calculated for the intervention group pre intervention and 2 weeks post intervention (case) and pre intervention and after a 2 week waiting period for the Wait Group (Control).
Time Frame: 2 weeks- 1 month
Population: medical students
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Wait Group | Intervention
Number analyzed (Participants) | 29 | 34
change in score on a scale | -0.52 (2.25) | -0.47 (2.34)
Statistical Analysis 1: Comparison: Wait Group vs Intervention; Test type: Superiority; p = .468104, t-test, 2 sided; The groups were compared using a two tailed unpaired t test with 61 degrees of freedom

ADVERSE EVENTS:
Time Frame: Adverse event information was collected over the course of the study and for 1 month after, so 3 months total.
Arm/Group | Intervention | Wait Group
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/29
Other Adverse Events (participants affected / at risk) | 0/34 | 0/29

LIMITATIONS AND CAVEATS:
The study period was brief, to stay within the timeframe of the Small Business Innovation Research (SBIR) Phase II grant. Additional follow-up time and intervention use would be needed to fully assess the impact of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT04494633/Prot_SAP_000.pdf